CLINICAL TRIAL: NCT02588235
Title: Impact of Combined Ezetimibe and Atorvastatin Therapy on Coronary Thin-cap Fibroatheroma As Assessed by Optical Coherence Tomography
Brief Title: Ezetimibe and Atorvastatin Therapy on TCFA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, sunddong, Attending, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TCFA-OCT XIJING01
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ezetimibe; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ezetimibe and Atorvastatin Therapy (Experimental): Atorvastatin (20 mg/day）plus ezetimibe（10 mg/day）
  Interventions: Drug: Ezetimibe and Atorvastatin
- Atorvastatin Therapy (Active Comparator): Atorvastatin (20 mg/day）
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Ezetimibe and Atorvastatin — atorvastatin (20 mg/day）plus ezetimibe（10 mg/day）
  Other Names: Ezetrol and lipitor
  Arms: Ezetimibe and Atorvastatin Therapy
Drug: Atorvastatin — atorvastatin (20 mg/day）
  Other Names: Lipitor
  Arms: Atorvastatin Therapy

SUMMARY:
After successful coronary angiography and OCT examination, patients with TCFAs in non-culprit, mild-to-moderate stenotic lesions will be enrolled. Then, they will be randomly assigned in a 1:1 ratio to receive either atorvastatin (20 mg/day) alone or atorvastatin (20 mg/day）plus ezetimibe（10 mg/day）by envelope method. Angiographic and OCT follow-up will be scheduled for the target vessel after 12 months.

DETAILED DESCRIPTION:
This is a prospective, randomized , controlled, open-label, single-center study to evaluate the effect of ezetimibe added to atorvastatin on coronary thin-cap fibroatheroma(TCFA). After successful coronary angiography and OCT examination, patients with TCFAs in non-culprit, mild-to-moderate stenotic lesions will be enrolled. Then, they will be randomly assigned in a 1:1 ratio to receive either atorvastatin (20 mg/day) alone or atorvastatin (20 mg/day）plus ezetimibe（10 mg/day）by envelope method.

Angiographic and OCT follow-up will be scheduled for the target vessel after 12 months.The primary efficacy endpoint is the change in minimum fibrous cap thickness measured by OCT from baseline to follow-up.The secondary endpoints include absolute and percent changes in the lipid, glycemic, and inflammatory profile. Then, changes of these indicators above will be compared respectively in diabetic and non-diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1.stable angina or acute coronary syndrome 2.18-80 years old 3.hypercholesterolemia :total cholesterol level >220 mg/dl (5.7mmol/L) and/or LDL-C level >140 mg/dl(3.6mmol/L), or previously receiving statins therapy 4. the target vessel for OCT interrogation has not undergone angioplasty and has angiographic diameter stenosis from 25% to 75% 5.There are TCFAs in non-culprit, mild-to-moderate stenotic lesions above

Exclusion Criteria:

1. administration of lipid-lowering drugs other than statins before enrollment
2. significant stenotic lesions in all coronary vessels
3. severe congestive heart failure (New York Heart Association class IV) ,or left ventricular ejection fraction<35%
4. more than 3 times of the upper limit of normal (ULN) in the creatine kinase (CK) and the transaminase level before enrollment and no relation with myocardial infarction
5. renal failure (serum creatinine>2.0 mg/dL）
6. hypersensitivity to x-ray contrast media, statin，clopidogrel or ezetimibe
7. Others: terminal stage cancer,a positive pregnancy test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
minimum fibrous cap thickness | 12months
  The primary efficacy endpoint is the change in minimum fibrous cap thickness measured by OCT from baseline to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, M.D., Ph.D., Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China